CLINICAL TRIAL: NCT02782195
Title: Validation of the Gut Absorption Rate of Glucose During a Large, Slowly and Rapidly-absorbed Evening Meal in Subjects With Type 1 Diabetes
Brief Title: Evaluation of Gut Absorption Rate of Glucose After a Large Evening Meal in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David Dunger, Professor of Paediatrics, University of Cambridge
Other Study IDs: APCam04
Record Dates: First submitted 2015-12-17; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Eight adolescent and young adult subjects with type 1 diabetes, age 16-24 years, will be recruited for this study on the basis of informed consent. Participants will be invited to attend the Wellcome Trust Clinical Research Facility at Addenbrooke's Hospital, Cambridge, on two occasions. On each occasion participants will arrive at the unit at 9am having controlled their diabetes with short acting insulin for 24 hours and they will remain in the unit until 8am the next morning. During the day, between 9am and 6pm participants will remain fasting and their blood glucose levels will be controlled by intravenous insulin, the dose being determined by 15-30 minute blood glucose estimations. At 1800hr on visit 1 the subjects will be asked to ingest an evening meal enriched by a cold isotope glucose tracer (non radioactive). The variable insulin infusion will be adjusted to allow for the meal in order to achieve good glycaemic control after the meal until 0200hr. From then until 0800hr in the morning the study team will again adjust the infusion rates to maintain normal glycemia until the participants are ready to go home on their normal insulin regimen. On the second visit the protocol will be identical until 1800hr when instead of giving the meal variable amounts of glucose will be infused to ensure the glucose levels are identical to those observed on visit 1. After 0200hr the study will be effectively finished but the study team will continue to vary the insulin infusion to keep blood glucose levels normal until the subjects can go home on their normal insulin regime at 8am.

In order to achieve sufficient information to make all the calculations needed other cold isotope glucose tracers will be infused during the study period. These safe non radioactive isotope tracers will enable us to assess glucose being produced by the body, its distribution and utilization. Throughout both study periods the subjects will be monitored very closely by a Clinical Research Fellow, assisted by a Research Nurse, in order to avoid any risk of low blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 16 and 24 years of age (inclusive)
* The subject has type 1 diabetes, as defined by WHO for at least 6 months or is confirmed C-peptide negative
* The subject will have been on insulin pump or MDI therapy for at least 6 months
* Body Mass Index (BMI) < 30 kg/m2
* HbA1c ≤ 12 % based on analysis from central laboratory

Exclusion Criteria:

* Non-type 1 diabetes mellitus including those secondary to chronic disease
* Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results
* Current treatment with drugs known to interfere with glucose metabolism such as systemic corticosteroids, non-selective beta-blockers and MAO inhibitors
* Experienced recurrent severe hypoglycaemic unawareness (as judged by the investigator)
* Known or suspected allergy against insulin
* Subjects with clinical significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator.
* Total daily insulin dose = 1.4 IU/kg.
* Pregnancy or intention of becoming pregnant, breast-feeding or judged to be using inadequate contraceptive methods. Adequate contraceptive methods are sterilisation, intrauterine device (IUD), oral contraceptives or consistent use of barrier methods
* Gastroparesis
* Symptomatic hypoglycaemia within 48h prior to study nights
* Moderate or intense exercise within 24h prior to study nights

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young adults with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To measure the rate of glucose absorption after a standard evening meal | Through study completion, up to 2 years, from date of randomization until the date of completion of data analysis
  Validation of the rate of glucose absorption after a large, slowly and rapidly-absorbed evening meal in subjects with type 1 diabetes.